CLINICAL TRIAL: NCT03574337
Title: Residual Neuromuscular Blockade in Cardiac Surgery Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mary Jarzebowski, Anesthesiologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Henryford
Record Dates: First submitted 2018-05-28; First posted 2018-07-02 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Residual neuromuscular blockade; Reversal; Cardiac surgery
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sugammadex (Active Comparator): Patient's will receive sugammadex at the end of the case for reversal of neuromuscular blockade. The dosing will be determined based on the patient's weight and TOF ratio by the pharmacy. It will be a one time dose at the end of the case
  Interventions: Drug: Sugammadex
- Neostigmine/glycopyrrolate (Active Comparator): Patient's will receive neostigmine/glycopyrrolate at the end of the case for reversal of neuromuscular blockade. The dosing will be determined based on the patient's weight (50mcg/kg of neostigmine with an equivalent volume to volume ratio of glycopyrrolate). It will be a one time dose at the end of the case
  Interventions: Drug: neostigmine/glycopyrolate
- No reversal administered (No Intervention): No reversal administered at the end of the case

INTERVENTIONS:
Drug: Sugammadex — No additional information
  Arms: Sugammadex
Drug: neostigmine/glycopyrolate — No additional information
  Arms: Neostigmine/glycopyrrolate

SUMMARY:
The purpose of this project is to determine if reversal of neuromuscular blockade in cardiac surgery patients expedites time to extubation in fast track patients.

DETAILED DESCRIPTION:
Neuromuscular blocking agents are used as part of most general anesthetics to help facilitate tracheal intubation and optimal surgical conditions (Barish et al). These medications cause universal paralysis of patients while unconscious. After most surgeries where extubation is planned, the standard of care is to "reverse" any residual neuromuscular blockade with either anticholinesterase treatment (specifically neostigmine) or sugammadex. Despite adequate reversal, residual neuromuscular blockade is a common problem seen in the post-anesthetic care unit (PACU). It leads to issues of airway obstruction, hypoxemia, respiratory complications including atelectasis and pneumonia and muscle weakness (Brull et al). The investigators posit that these complications are likely amplified in patients who require post-operative intensive care unit admission. In particular, the investigators hypothesize that cardiac surgery patients are at risk. Elective cardiac surgery patients are routinely admitted to the CVICU still intubated and ventilator-dependent immediately following surgery. The goal of uncomplicated cardiac surgery patients (fast track cardiac surgery patients) is to extubate them within 6 hours of ICU arrival. However, standard of care throughout the US does not include reversal of their neuromuscular blockade. By the time these patients meet extubation criteria, most providers believe that the neuromuscular blockade should have worn off and therefore do not administer reversal (Murphy et al). The investigators hypothesize that residual neuromuscular blockade delays time to extubation and increases respiratory complications in fast track cardiac surgery patients. By administering reversal of neuromuscular blockade in patients with a Train Of Four ratio of <0.9 we anticipate that there will be an increase from 60 to 85% of patients being successfully extubated within 6 hours of arrival to the ICU and a decrease in composite respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients >18 years of age scheduled for elective coronary artery bypass graft surgery (CABG), aortic valve replacement (AVR), or combination CABG/AVR

Exclusion Criteria:

* Chronic kidney disease stage IV or V
* Liver disease, defined as AST, ALT or ALP > 1.5x upper limit of normal Inpatient status
* Allergy to rocuronium

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Time from arrival in CVICU until extubation | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Tidal volumes prior to extubation | Prior to extubation, the tidal volumes the patient is generating will be documented
Need for unplanned noninvasive positive pressure ventilation or high flow nasal cannula | through study completion, an average of 1 year
  Assess how many liters of oxygen the patient requires to maintain pulse oximetry >92%
Lowest documented pulse oximetry | through study completion, an average of 1 year
Number of participants requiring re-intubation | through study completion, an average of 1 year
  If the patient is extubated in the intensive care unit but then develops respiratory failure and requires mechanical ventilation again
Bronchoscopy | through study completion, an average of 1 year
  Change in baseline oxygen requirements from prior to the surgery
Pneumonia | through study completion, an average of 1 year
  Change in baseline oxygen requirements from prior to the surgery
Intensive care unit length of stay | through study completion, an average of 1 year
Mortality | 28 days following the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jarzebowski, MD, Principal Investigator — Henry Ford Health Systems
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu F, Lee A, Chee YE. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2012 Oct 17;10:CD003587. doi: 10.1002/14651858.CD003587.pub2. PMID 23076899
- [Result] Richey M, Mann A, He J, Daon E, Wirtz K, Dalton A, Flynn BC. Implementation of an Early Extubation Protocol in Cardiac Surgical Patients Decreased Ventilator Time But Not Intensive Care Unit or Hospital Length of Stay. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):739-744. doi: 10.1053/j.jvca.2017.11.007. Epub 2017 Nov 8. PMID 29229252